CLINICAL TRIAL: NCT01971801
Title: Vitamin D Supplementation in Older Adults With Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alayne D. Markland, DO, MSc, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAMC11
Record Dates: First submitted 2013-10-17; First posted 2013-10-29 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Urinary Incontinence; Vitamin D Deficiency
Keywords: urinary incontinence; bowel incontinence; vitamin D; overactive bladder; lower urinary tract symptoms; quality of life
MeSH Terms: conditions — Urinary Incontinence; Vitamin D Deficiency; Fecal Incontinence; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D3, 50,000 IU, weekly
  Interventions: Dietary Supplement: Vitamin D3 50,000 IU
- Placebo (Placebo Comparator): Placebo comparator, weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 50,000 IU — Capsule given by mouth once a week
  Arms: Vitamin D
Other: Placebo — One capsule given by mouth weekly
  Other Names: Capsule placebo
  Arms: Placebo

SUMMARY:
Urinary incontinence (UI) is a common disorder among older women that greatly affects quality of life. Emerging evidence from observational studies links vitamin D insufficiency with UI. Prior to a larger intervention trial of vitamin D among older women with low serum vitamin D levels and urgency UI, we propose a pilot study in 100 older women comparing weekly, oral vitamin D3 50,000 IU to placebo. We hypothesize that adequate vitamin D supplementation will improve UI symptoms in older women with vitamin D deficiency. Changes in UI-episodes will be assessed by a 7-day bladder diary and other validated symptom measures administered at baseline and after 12-weeks of intervention. Serum calcium and 25(OH)D levels will be monitored. The expected outcomes will provide new knowledge regarding the impact of vitamin D supplementation on UI symptom improvement and inform a larger, randomized controlled clinical trial involving vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

(1) Post-menopausal women (age ≥50 years of age); (2)Urine leakage for 3 or more months; (3) at least 3 urinary urgency incontinence episodes on a 7-day bladder diary; and (4) serum 25(OH)D level (vitamin D) is <30 ng/mL. Women who currently take a bladder medications (anticholinergic) for UI symptom control may enroll into the study if they agree to (1) cease taking these medications at least two weeks before the pre-intervention assessment and (2) not take these medications during the study's treatment and assessment period.

Exclusion Criteria:

(1) neurologic diseases known to affect UI; (2) Diseases known to affect vitamin D absorption and metabolism; (3) Prior pelvic floor radiation; (4) Obstructive causes of UI;(6)Current use of medications known to affect vitamin D levels; (7) Uncontrolled diabetes (Hemoglobin A1C>9%); (8) albumin corrected serum Calcium > 11.0 mg/dL; (9)history of hyperparathyroidism; (10) currently untreated kidney stones; (11) post void residual urine volume >200 ml; and, (12) current treatment with vitamin D >=1000IU/day (if not willing to stop taking).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in the number of incontinent episodes on a 7-day bladder diary | baseline to 12 weeks
  The primary outcome measure is the percentage change in the number of incontinent episodes on a 7-day bladder diary from the baseline evaluation to the final visit at 12-weeks.

SECONDARY OUTCOMES:
Change in UI symptoms (ICIQ-UI and ICIQ-OAB scores) | baseline to 12 weeks
  Questionnaires
Change in quality of life (Overactive Bladder Questionnaire) | baseline to 12 weeks
  Questionnaires
Change in satisfaction with treatment (Perceptions and Satisfaction Questionnaire) | baseline to 12 weeks
  Questionnaire
Change in safety of the treatments (side effects and unanticipated events) | baseline to 12 weeks
  Checklist
Mechanisms of improvement based on measure of mobility | baseline to 12 weeks
  Physical examination
Bowel incontinence symptoms | baseline to 12 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alayne D Markland, DO, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Continence Clinic at The Kirklin Clinic, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Markland AD, Tangpricha V, Mark Beasley T, Vaughan CP, Richter HE, Burgio KL, Goode PS. Comparing Vitamin D Supplementation Versus Placebo for Urgency Urinary Incontinence: A Pilot Study. J Am Geriatr Soc. 2019 Mar;67(3):570-575. doi: 10.1111/jgs.15711. Epub 2018 Dec 21. PMID 30578542